CLINICAL TRIAL: NCT03354728
Title: A Phase 1/2 Clinical Study to Evaluate the Optimal Dose and the Protective Effect of CMV-MVA Triplex Vaccine in Pediatric Patients Receiving an Allogeneic Hematopoietic Stem Cell Transplant
Brief Title: Multi-antigen CMV-Modified Vaccinia Ankara Vaccine in Treating Pediatric Patients With Positive Cytomegalovirus Undergoing Donor Stem Cell Transplant
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17236; NCI-2017-02046 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17236 (Other: City of Hope Comprehensive Cancer Center)
Record Dates: First submitted 2017-11-06; First posted 2017-11-28 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Cytomegaloviral Infection; Hematopoietic Cell Transplant Recipient
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive Care (multi-antigen CMV-modified vaccinia ankara) (Experimental): Patients receive multi-antigen CMV-modified vaccinia ankara vaccine IM on days 28 and 56 post-HCT.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Multi-peptide CMV-Modified Vaccinia Ankara Vaccine

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Multi-peptide CMV-Modified Vaccinia Ankara Vaccine — Given IM
  Other Names: CMV-MVA Triplex Vaccine; Multi-antigen CMV-Modified Vaccinia Ankara Vaccine

SUMMARY:
This phase I/II trial studies the side effects and best dose of multi-antigen cytomegalovirus (CMV)-modified vaccinia ankara vaccine and to see how well it works in treating pediatric patients with positive cytomegalovirus who are undergoing donor stem cell transplant. Multi-antigen CMV-modified vaccinia ankara vaccine may help people resist CMV life-threatening complications.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate the optimal dose of multi-antigen CMV-modified vaccinia ankara vaccine (Triplex) in CMV-positive pediatric patients receiving human leukocyte antigen (HLA) matched, mismatched, or haploid-identical hematopoietic cell transplantation (HCT). (Phase I) II. To evaluate the safety profile of Triplex in this patient population. (Phase I) III. To determine if Triplex reduces the frequency of CMV events when compared to historical data. (Phase II)

SECONDARY OBJECTIVES:

I. To characterize CMV reactivation and disease by assessing: time to CMV reactivation, duration of viremia, recurrence of viremia, incidence of late CMV viremia/disease (defined as > 100 days and =< 365 days post HCT), use of anti-viral drugs triggered by rising CMV viremia or viremia >= 3750 IU/mL, cumulative number of CMV specific antiviral treatment days.

II. To evaluate the impact of Triplex on transplant related outcomes by assessing the incidence of acute and chronic graft versus host disease (GVHD), relapse, non-relapse mortality (NRM), all-cause mortality, infections.

III. To investigate the impact of Triplex on cellular immunity by investigating: the level, function and kinetics of CMV-specific T-cell immunity, the changes in adaptive natural killer (NK) cell population and highly cytotoxic memory NKG2C+ NK cells, and changes in GVHD biomarkers.

OUTLINE: This is a phase I, dose-escalation study followed by a phase II study.

Patients receive multi-antigen CMV-modified vaccinia ankara vaccine intramuscularly (IM) on days 28 and 56 post-HCT.

After completion of study treatment, patients are followed up for up to 270 or 365 days.

ELIGIBILITY:
Inclusion Criteria:

* All subjects (or their guardians) must have the ability to understand and the willingness to sign a written informed consent; age appropriate assent will be obtained per institutional guidelines; to allow non-English patients to participate in this study, bilingual health services will be provided in the appropriate language when feasible
* Participant must be willing to comply with study and/or follow-up procedures, including willingness to be followed for one year post-HCT
* Planned allogenic (allo)-HCT, with 9/10 or 10/10 (A, B, C, DRB1, DQB1) high/intermediate resolution HLA donor allele matching and with no T-cell depletion of graft
* Planned related HCT with molecular 3/6 HLA donor allele matching (haploidentical) (for phase I only)
* CMV seropositive at the time of HCT
* Conditioning and immunosuppressive regimens according to institutional guidelines are permitted
* Negative serum or urine beta-human chorionic gonadotropin (HCG) test (female patient of childbearing potential only) within two weeks of registration
* Seronegative for human immunodeficiency virus (HIV), hepatitis C virus (HCV); if hepatitis B virus (HBV) core seropositive, absence of HBV deoxyribonucleic acid (DNA) within 2 months of registration
* Agreement by females of childbearing potential and sexually active males to use an effective method of contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for up to 90 days post-HCT; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately

Exclusion Criteria:

* TRANSPLANT RELATED CRITERIA: Patients undergoing cord blood transplant (CB-HCT)
* Any prior investigational CMV vaccine
* Anti-CMV therapy in the last 6 months
* Live attenuated vaccines
* Medically indicated subunit (Engerix-B for HBV; Gardasil for human papillomavirus [HPV]) or killed vaccine (e.g. influenza, pneumococcal)
* Allergy treatment with antigens injections
* Alemtuzumab, cyclophosphamide, ATG or any equivalent in vivo T-cell depleting agent; Note: Pre-transplant ATG is permitted
* Antiviral medications with known therapeutic effects on CMV such as ganciclovir (GCV)/valine (VAL), FOS, Cidofovir, CMX-001, maribavir; acyclovir has no known therapeutic efficacy against CMV and is allowable as standard of care to prevent herpes simplex virus (HSV)
* Prophylactic therapy with CMV immunoglobulin or prophylactic antiviral CMV treatment; intravenous immunoglobulin therapy (IVIG) is allowed
* Other investigational product-concurrent enrollment in other clinical trials using any investigational new drug (IND) drugs with unknown effects on CMV or with unknown toxicity profiles is prohibited
* Other medications that might interfere with the evaluation of the investigational product
* Patients with congenital immune deficiency
* Patients with active autoimmune conditions requiring systemic immunosuppressive therapy within the previous 5 years are not eligible, the exception to this is patients with aplastic anemia, who are eligible
* Pregnant women and women who are lactating; CMV-MVA Triplex risks to pregnant women are unknown; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with the administered vaccine, also breastfeeding should be discontinued if the mother is enrolled on this study
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., social/psychological issues, etc
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issue related to feasibility/logistics)

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-05-11 (Actual); Primary Completion 2026-12-11 (Estimated); Study Completion 2026-12-11 (Estimated)

PRIMARY OUTCOMES:
Optimal dose (Phase I) | Up to 1 year
Incidence of adverse events (Phase I) | Up to 1 year
  Adverse events will be characterized using the descriptions and grading scales according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Cytomegalovirus (CMV) events (reactivation >= 1250 IU/mL), or viremia treated by anti-viral therapy, or detection of CMV by histology (Phase II) | Prior to day 100 post-hematopoietic cell transplantation (HCT) or viremia treated by anti-viral therapy, or detection of CMV by histology
  Will be assessed with exact 90% confidence bounds.
Non-relapse mortality | At 100 days post-HCT
  Will be compared to historical controls at the final analysis, and a 90% lower confidence bound on the difference in 12-month event free survival will be produced.
Severe (grade 3-4) acute graft versus host disease (aGVHD) | Within 2 weeks from each vaccination
Incidence of grade 3-4 adverse events | Within 2 weeks from each vaccination
  Will be graded per CTCAE version 4.0.

SECONDARY OUTCOMES:
Time-to viremia | Number of days from transplant to the date of > 1250 IU/mL, assessed up to 1 year
Duration of viremia | Up to 1 year
Incidence of late CMV viremia | > 100 and =< 365 days post-HCT
Use of antiviral drugs (triggered by rising CMV viremia or viremia >= 3,750 IU/ml) | Up to 1 year, rising CMV viremia or viremia >= 3,705
Cumulative number of CMV specific antiviral treatment days | Up to 1 year
Time to engraftment | Up to 1 year
Incidence of acute graft versus host disease (aGVHD) | Up to 1 year
Chronic GVHD (cGVHD) | Up to 1 year
Relapse defined by bone marrow and/or imaging studies | Up to 1 year
Non-relapse mortality | Up to 1 year
All-cause mortality | Up to 1 year
Infections | Up to 1 year
Levels of CMV-specific T cell immunity | Up to 1 year post-HCT
  Will be combined with immunophenotyping and functional studies. The data analysis for estimating the effect of vaccination on cellular immunity will necessarily be more exploratory in nature. The longitudinal CMV-specific cellular assay data will be modeled on a logarithmic scale, using a generalized estimating equation approach to accommodate the stochastic dependence through time. This produces an estimated multiplicative effect of vaccination, qualified by a valid estimate of variability.
Kinetics of CMV-specific T cell immunity | Up to 1 year post-HCT
  The data analysis for estimating the effect of vaccination on cellular immunity will necessarily be more exploratory in nature. The longitudinal CMV-specific cellular assay data will be modeled on a logarithmic scale, using a generalized estimating equation approach to accommodate the stochastic dependence through time. This produces an estimated multiplicative effect of vaccination, qualified by a valid estimate of variability.
Natural killer (NK) phenotype | Up to 1 year post-HCT
  The data analysis for estimating the effect of vaccination on cellular immunity will necessarily be more exploratory in nature. The longitudinal CMV-specific cellular assay data will be modeled on a logarithmic scale.
NK function (cytotoxicity and cytokine production) | Up to 1 year post-HCT
  The data analysis for estimating the effect of vaccination on cellular immunity will necessarily be more exploratory in nature. The longitudinal CMV-specific cellular assay data will be modeled on a logarithmic scale, using a generalized estimating equation approach to accommodate the stochastic dependence through time. This produces an estimated multiplicative effect of vaccination, qualified by a valid estimate of variability.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Pawlowska, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States